CLINICAL TRIAL: NCT05043766
Title: A Phase 1b, Randomized 2-Part Single-Center Study to Evaluate the PK and Safety of Multiple Ascending Oral Doses of PF614 and the Food Effect and BA/BE of Single Oral Doses of PF614 Relative to OxyContin in Healthy Adult Subjects
Brief Title: Evaluation of Oral PF614 Relative to OxyContin (PF614-102)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ensysce Biosciences (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PF614-102
Record Dates: First submitted 2021-09-02; First posted 2021-09-14 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Healthy Volunteers
Keywords: Prodrug; PF614; OxyContin; oral
MeSH Terms: interventions — Naltrexone; Oxycodone

STUDY DESIGN:
Intervention Model Description: Part A will utilize a randomized, open label, multiple-ascending dose design with up to 3 separate dose groups of 8 subjects per group.
  Part B will utilize an open-label, single-dose, randomized, 4-way crossover design with 13 subjects in each treatment sequence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PF614 (Experimental): Part A will utilize a randomized, open-label, multiple-ascending dose design with up to 3 separate dose groups of 8 subjects. Within each dose group, subjects will be randomized to receive repeated BID doses, planned to be 12 hours apart over a 5 day period, for a total of 9 doses. Dose escalation to Dose Groups 2 and 3 will follow a review of pharmacokinetic, safety and tolerability data up to Day 10 of the preceding group. The doses or dosing regimen for Dose groups 2 and 3 may be modified based on a review of the data.
  Interventions: Drug: PF614; Drug: Naltrexone Hydrochloride
- Part B Compare Bioavailability and Bioequivalence (Active Comparator): Part B will utilize an open-label, single-dose, randomized, 4-way crossover design. Following confirmation of eligibility, subjects will be randomized to receive each of the single oral doses of study drugs (one at each treatment period).
  PF614 100 mg administered under fasted conditions; PF614 100 mg administered under fed conditions; OxyContin 40 mg administered under fasted conditions; OxyContin 40 mg administered under fed conditions
  Interventions: Drug: PF614; Drug: Naltrexone Hydrochloride; Drug: OxyContin

INTERVENTIONS:
Drug: PF614 — PF614 is an oxycodone prodrug
  Other Names: oxycodone prodrug
Drug: Naltrexone Hydrochloride — Naltrexone HCl tablets, 50 mg, will be used to block the opioid effects in healthy volunteers
  Other Names: ReVia
Drug: OxyContin — Bioequivalence single-dose comparison to OxyContin
  Other Names: OxyContin 40 mg Extended-Release Tablet
  Arms: Part B Compare Bioavailability and Bioequivalence

SUMMARY:
This is a single-center study incorporating 2 parts: A Multiple Ascending Dose Study (Part A) and a comparative Bioavailability/Bioequivalence and Food Effect study (Part B). Both parts of the study will be conducted in healthy adult subjects.

DETAILED DESCRIPTION:
This study is intended to evaluate the pharmacokinetics of OxyContin (oxycodone ER) and PF614, as well as PF614 fragments, following administration of multiple ascending doses of PF614, and to compare to steady-state pharmacokinetics to those of OxyContin. (Part A)

In addition, oral bioavailability of oxycodone derived from single doses of PF614 of the to-be-marketed capsule formulation will be compared to that of the reference drug, OxyContin, in the fasted and fed condition. A pivotal food effect assessment will be incorporated into the study to determine the impact of a high fat meal on the bioavailability of oxycodone, following oral single-dose administration of PF614 (Part B).

ELIGIBILITY:
Inclusion Criteria:

* Males or females, ages 18-50 years in good general health,
* BMI between 18 and 32 kg/m (inclusive)
* Subjects must have a negative screen for drugs of abuse, nicotine, alcohol, Hepatitis B, Hepatitis C, and HIV.
* Female subjects of child bearing potential must have a negative serum pregnancy test at randomization
* Females must be of non-child bearing potential (e.g. postmenopausal) or of childbearing potential and agree to use a highly effective form of contraception from the time of screening to two weeks after last dose of study medication.
* Subjects must have normal findings in a physical examination and 12 lead ECG and normal Vital Signs
* Clinical laboratory values must be Within Normal limits as defined by the clinical laboratory
* Subjects must be able to provide coherent written informed consent
* Subjects must be willing and able to follow study instructions and be likely to complete all study requirements.

Exclusion Criteria:

* History of allergy or sensitivity to oxycodone
* History of loud snoring or sleep apnea
* History of medical problems encountered with opioid therapy
* Urinary cotinine levels indicative of smoking or history of smoking or regular tobacco use with 2 months prior to screening
* History of alcoholism or drug abuse
* Use of prescription medications within 14 days of study drug administration with exception of contraceptives used by female subjects
* Use of any opioid within 30 days prior to screening
* History of allergy or sensitivity to naltrexone
* History of allergy or sensitivity to naloxone
* Donation of blood within 30 days prior to screening
* Donation of plasma within 30 days prior to screening
* Acute illness at admission of clinical study unit
* History of GI disturbance requiring use of antacid twice weekly or more
* Females who are breastfeeding
* Anticipated need for surgery or hospitalization during the study
* Enrollment in an investigational drug study within 30 days prior to screening
* Any condition that in the Investigator's opinion puts the subject at significant risk, could confound the study results, or may interfere significantly with the subject's participation in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 30 days
  Adverse Events, Significant Adverse Events, Adverse Events leading to discontinuation
Pharmacokinetics AUC [Area Under the Curve] | Full PK sampling time points will be 0, 30 minutes; 1, 2, 3, 4, 6, 8, and 12 hours
  Area under the concentration-time curve from the time of dosing to the start of the next dosing interval using PF614 concentrations and oxycodone concentrations in plasma.
Pharmacokinetics Cmax [Maximum Plasma Concentration] | PK sampling time points will be 0, 30 minutes; 1, 2, 3, 4, 6, 8, and 12 hours
  Maximum (peak) plasma concentration first dose
Pharmacokinetics Tlag [Time to first measurable plasma concentration] | PK sampling time points will be 0, 30 minutes; 1, 2, 3, 4, 6, 8, and 12 hours
  Time prior to the time corresponding to the first measurable (non-zero) concentration
Pharmacokinetics Tmax [Time to maximum plasma concentration] | PK sampling time points 30 minutes; 1, 2, 3, 4, 6, 8, and 12 hours
  Time to maximum plasma concentration on Day 1 (first dose)
Pharmacokinetics AUC, Steady State | PK sampling time points 0, 30 minutes; 1, 2, 3, 4, 6, 8, and 12 hours
  Steady-state (Day 5) area under the concentration-time curve from the time of dosing extrapolated to time infinity
Pharmacokinetics CL/F [Clearance] | PK sampling time points 0, 30 minutes; 1, 2, 3, 4, 6, 8, and 12 hours
  Apparent total systemic clearance
Pharmacokinetics Cmax, Steady State | PK sampling time points 0, 30 minutes; 1, 2, 3, 4, 6, 8, and 12 hours
  Maximum (peak) plasma concentration at steady-state on Day 5
Pharmacokinetics Tmax, Steady State | PK sampling time points 0, 30 minutes; 1, 2, 3, 4, 6, 8, and 12 hours
  Time to maximum plasma concentration on Day 5
Pharmacokinetics t1/2 [Half-life] | PK sampling time points 0, 30 minutes; 1, 2, 3, 4, 6, 8, and 12 hours
  Terminal elimination half-life
Pharmacokinetics Vz/F [Volume of Distribution] | PK sampling time points 0, 30 minutes; 1, 2, 3, 4, 6, 8, and 12 hours
  Apparent volume of distribution during the terminal-elimination phase
Pharmacokinetics elimination rate | PK sampling time points 0, 30 minutes; 1, 2, 3, 4, 6, 8, and 12 hours
  Terminal elimination rate/constant
Pharmacokinetics Ctrough [Minimum Plasma Concentration before next dose] | Prior to dosing on Days 2, 3, and 4
  Concentrations prior to dosing
Pharmacokinetics Part B AUC | PK sampling time points 0, 30 minutes; 1, 2, 3, 4, 6, 8, and 12 hours
  Area under the concentration-time curve from the time of dosing extrapolated to time infinity in fed vs fasted state
Pharmacokinetics Part B AUC 0-t | PK sampling time points 0, 30 minutes; 1, 2, 3, 4, 6, 8, and 12 hours
  Area under the concentration-time curve from the time of dosing to the last measurable concentration in fed vs fasted state
Pharmacokinetics Part B Cmax | PK sampling time points 0, 30 minutes; 1, 2, 3, 4, 6, 8, and 12 hours
  Maximum (peak) plasma concentration in fed vs fasted state
Bioavailability and Bioequivalence | PK sampling time points 0, 30 minutes; 1, 2, 3, 4, 6, 8, and 12 hours
  Bioavailability and Bioequivalence of single oral doses of PF614 prodrug and oxycodone derived from from PF614 vs. oxycodone derived from OxyContin in healthy adult subjects (Part B)

SECONDARY OUTCOMES:
Pharmacokinetics Part B CL/F | PK sampling time points 0, 30 minutes; 1, 2, 3, 4, 6, 8, and 12 hours
  Apparent total systemic clearance
Pharmacokinetics Part B pAUC | PK sampling time points 0, 30 minutes; 1, 2, 3, 4, 6, 8, and 12 hours
  Partial area under the concentration-time curve from the time of dosing to 12 hours post dose
Pharmacokinetics Part B Tlag | PK sampling time points 0, 30 minutes; 1, 2, 3, 4, 6, 8, and 12 hours
  Time prior to the time corresponding to the first measurable dose (non-zero) concentration
Pharmacokinetics Part B Tmax | PK sampling time points 0, 30 minutes; 1, 2, 3, 4, 6, 8, and 12 hours
  Time to maximum plasma concentration on Day 1 (first dose)
Pharmacokinetics Part B t1/2 | PK sampling time points 0, 30 minutes; 1, 2, 3, 4, 6, 8, and 12 hours
  Terminal elimination half life
Pharmacokinetics Part B Vz/F | PK sampling time points 0, 30 minutes; 1, 2, 3, 4, 6, 8, and 12 hours
  Apparent volume of distribution during the terminal elimination phase
Pharmacokinetics Part B Terminal elimination rate | PK sampling time points 0, 30 minutes; 1, 2, 3, 4, 6, 8, and 12 hours
  Terminal elimination rate constant
Plasma Concentration of inactive metabolic fragment #1 | PK sampling time points 0, 30 minutes; 1, 2, 3, 4, 6, 8, and 12 hours
  Evaluate plasma concentrations of PFR06082 (Part A only)
Plasma Concentration of inactive metabolic fragment #2 | PK sampling time points 0, 30 minutes; 1, 2, 3, 4, 6, 8, and 12 hours
  Evaluate plasma concentrations of PFR06110 (Part A only)

CONTACTS AND LOCATIONS:
Overall Officials: William K Schmidt, PhD, Study Director — Chief Medical Officer, Ensysce Biosciences
Locations (1):
- PRA Health Sciences-Early Development Services, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirkpatrick DL, Evans C, Pestano LA, Millard J, Johnston M, Mick E, Schmidt WK. Clinical evaluation of PF614, a novel TAAP prodrug of oxycodone, versus OxyContin in a multi-ascending dose study with a bioequivalence arm in healthy volunteers. Clin Transl Sci. 2024 Mar;17(3):e13765. doi: 10.1111/cts.13765. PMID 38511523
- [Background] Kirkpatrick DL, Schmidt WK, Morales R, Cremin J, Seroogy J, Husfeld C, Jenkins T. In vitro and in vivo assessment of the abuse potential of PF614, a novel BIO-MD prodrug of oxycodone. J Opioid Manag. 2017 Jan/Feb;13(1):39-49. doi: 10.5055/jom.2017.0366. PMID 28345745